CLINICAL TRIAL: NCT00306098
Title: Islet Cell Transplantation Alone in Patients With Type 1 Diabetes Mellitus: Steroid-Free Immunosuppression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rodolfo Alejandro (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Health Resources and Services Administration (HRSA) (U.S. Federal Agency); Diabetes Research Institute Foundation (Other); University of Miami (Other); National Center for Research Resources (NCRR) (NIH)
Responsible Party: Sponsor-Investigator, Rodolfo Alejandro, Professor of Medicine, University of Miami
Organization: University of Miami (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20000196; 1U42RR016603-01 (NIH); HRSA # 1 R38OT01367-01-00; No Number (Other Grant/Funding Number: Diabetes Research Institute Foundation, Miami Florida)
Record Dates: First submitted 2006-03-17; First posted 2006-03-22 (Estimated); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Diabetes Mellitus, Type I
Keywords: Transplantation, Islets of Langerhans
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Islets of Langerhans Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Islet transplantation (Experimental): Subjects receiving intraportal Islet cell infusion (transplant)
  Interventions: Drug: islets

INTERVENTIONS:
Drug: islets — Intraportal infusion of islets
  Other Names: islet transplantation

SUMMARY:
SPECIFIC AIMS:

1. To reverse hyperglycemia and insulin dependency in patients with Type 1 Diabetes Mellitus by islet cell transplantation;
2. To eliminate the incidence of hypoglycemia coma and unawareness in patients with Type 1 Diabetes Mellitus by islet cell transplantation;
3. To assess long-term safety and function of successful islet cell transplants in patients with Type 1 Diabetes Mellitus;
4. To determine whether the natural history of the microvascular, macrovascular and neuropathic complications of Diabetes Mellitus are altered following successful transplantation of islet cells; and
5. To assess the effect of infliximab in preventing early islet destruction, and thereby eliminating the need for a second donor's islet cells.
6. To assess the effect of etanercept in preventing early islet destruction.
7. To assess the effect of exenatide to improve islet graft function and survival in subjects that have returned to using exogenous insulin.
8. To assess the ability of exenatide to improve islet survival at time of transplantation.

DETAILED DESCRIPTION:
This Phase II trial will have 3 groups: Group A will receive islets from 2 donors and will not receive infliximab. Group B will receive, in addition to Daclizumab, Sirolimus, and Tacrolimus, a dose of infliximab and islets from a single donor, as per the Edmonton protocol. Everything else about the clinical trial will be the same for both groups. The first 4 patients will be assigned to Group A, the next 4 patients to Group B, the next 4 patients to Group A, and the next 4 patients to Group B (total =16). Patients in Group A will receive 1-2 transplants with cells from 2 donors. If the second donor pancreas is received and satisfactory at the same time as the first pancreas, one islet infusion will be used to infuse cells from both donors. If the second pancreas is not received until after the first transplantation, a second islet infusion will be done. A second course of five doses of Daclizumab will be started on the day of the second islet infusion).

In order to determine if prolonged administration of etanercept, in combination with transplantation of cultured islets, will prevent TNF-α production and enhance engraftment, we have added Group C to the current protocol. Group C, in addition to Daclizumab, Sirolimus, and Tacrolimus, will receive Etanercept in the peri-transplant period and islets from one or more donors. The last 24 patients included in this Protocol will be in Group C if they are new, or in Group A and B Supplemental Infusion if they had previous transplants. Any Group A or B participants who are eligible for a supplemental infusion will receive etanercept but no infliximab.

ELIGIBILITY:
Inclusion Criteria:

1. Patients between 18 and 65 years of age
2. Patients with type 1 diabetes mellitus for more than 5 years duration
3. One or more of the following:

   * Hypoglycemia unawareness - judged by history of blood sugars <54 on glucometer without symptoms and/or hypoglycemic episodes requiring assistance from either family, glucagon administration or emergency services
   * Poor diabetes control (HbA1c>8% or >2 visits/yr to hospital for treatment of ketoacidosis) despite intensive insulin therapy
   * Progressive complications of type 1 diabetes mellitus
4. Body Mass Index (BMI) ≤26

Exclusion Criteria:

1. c-peptide > 0.3ng/ml basal or stimulated;
2. untreated proliferative diabetic retinopathy;
3. HbA1C >12%;
4. creatinine clearance <60;
5. serum creatinine consistently >1.6 mg/dl;
6. macroalbuminuria >300mg albumin in 24 hours;
7. presence of panel reactive antibodies (PRA) >20%;
8. previous/concurrent organ transplantation (except previous unsuccessful islet cell transplant;
9. malignancy or previous malignancy (except non-melanomatous skin cancer);
10. x-ray evidence of pulmonary infection;
11. active infections;
12. active peptic ulcer disease, gall stones, hemangioma, or portal hypertension
13. serological evidence of HIV, HbsAg or HCV; serological evidence of active EBV (IgM>IgG) or EBV negative serology;
14. PPD conversion or positive PPD without historic completion of appropriate prophylactic treatment;
15. abnormal liver function test;
16. anemia (hemoglobin <12.0);
17. hyperlipidemia (fasting serum triglycerides >200mg/dl and/or fasting serum cholesterol >240 mg/dl and/or fasting LDL cholesterol >140 mg/dl);
18. BMI above 26;
19. unstable cardiovascular status; prostate specific antigen (PSA) >4;
20. pregnancy or breastfeeding;
21. sexually-active females who are not: a) post-menopausal, b) surgically sterile, or c) not using an acceptable method of contraception (oral contraceptives, Norplant, Depo-Provera, and barrier devices are acceptable; condoms used alone are not acceptable);
22. alcohol abuse, substance abuse or smoking within the previous 6 months; insulin requirement >1u/kg/day and any condition or any circumstance that makes it unsafe to undergo an islet cell transplant.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2000-12; Primary Completion 2004-07-04 (Actual); Study Completion 2004-07-04 (Actual)

PRIMARY OUTCOMES:
a1c less than 6.5 without severe hypoglycemia | for the duration of islet graft function
  number of subjects with a1c less than 6.5 without severe hypoglycemia

SECONDARY OUTCOMES:
partial graft function, as evidenced by baseline C-peptide greater than 0.5 ng/ml | 1 year
  Number of subjects with basal c-peptide greater than 0.5 ng/ml
reduction in insulin requirements in those patients who do not achieve insulin independence | 1 year
  Number of subjects with at least 40% reduction in insulin requirements
improvement in metabolic control as evidenced by improvement in: HbA1C (less or equal to 7) | 1 year
  Number of subjects with HBA1C less or equal to 7
elimination or reduction in the incidence of hypoglycemic coma or unawareness | 1 year
  Number of subjects without severe hypoglycemia
assessment of efficacy of infliximab in preventing early rejection - | 1 year
  number of subjects achieving insulin independence with a single infusion of infliximab vs no infliximab

CONTACTS AND LOCATIONS:
Overall Officials: Rodolfo Alejandro, M.D., Principal Investigator — University of Miami, Diabetes Research Institute; Camillo Ricordi, M.D., Principal Investigator — University of Miami, Diabetes Research Institute
Locations (1):
- University of Miami, Diabetes Research Institute, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Froud T, Ricordi C, Baidal DA, Hafiz MM, Ponte G, Cure P, Pileggi A, Poggioli R, Ichii H, Khan A, Ferreira JV, Pugliese A, Esquenazi VV, Kenyon NS, Alejandro R. Islet transplantation in type 1 diabetes mellitus using cultured islets and steroid-free immunosuppression: Miami experience. Am J Transplant. 2005 Aug;5(8):2037-46. doi: 10.1111/j.1600-6143.2005.00957.x. PMID 15996257
- [Derived] Faradji RN, Froud T, Messinger S, Monroy K, Pileggi A, Mineo D, Tharavanij T, Mendez AJ, Ricordi C, Alejandro R. Long-term metabolic and hormonal effects of exenatide on islet transplant recipients with allograft dysfunction. Cell Transplant. 2009;18(10):1247-59. doi: 10.3727/096368909X474456. PMID 20003758
- [Derived] Tharavanij T, Betancourt A, Messinger S, Cure P, Leitao CB, Baidal DA, Froud T, Ricordi C, Alejandro R. Improved long-term health-related quality of life after islet transplantation. Transplantation. 2008 Nov 15;86(9):1161-7. doi: 10.1097/TP.0b013e31818a7f45. PMID 19005394
- See also: Web site of Diabetes Research Institute, University of Miami — http://www.diabetesresearch.org